CLINICAL TRIAL: NCT05104632
Title: Financial Toxicity in Surgical Breast Cancer Patients: A Prospective, Multicenter Cohort Study
Brief Title: Financial Toxicity in Breast Cancer Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Juravinski Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 131916
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Financial toxicity; Breast cancer; Lumpectomy; Mastectomy; Breast reconstruction
MeSH Terms: conditions — Breast Neoplasms; Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast conserving surgery only: Patients who receive breast conserving surgery.
- Mastectomy only: Patients who receive mastectomy surgery.
- Mastectomy & breast reconstruction: Patients who receive mastectomy and breast reconstruction.

SUMMARY:
The purpose of this study is to evaluate financial toxicity, or financial harm, in breast cancer patients. The study will follow patients throughout their cancer treatment. The study investigators will measure if patients are experiencing financial toxicity and if it changes throughout treatment, and whether it's associated with different cancers, treatments, or demographics. Also, the study investigators will measure if financial toxicity impacts other areas of life (e.g., well-being, satisfaction). Finally, patients will be asked to estimate how much money they expect to spend on out-of-pocket expenses during their treatment and how their finances and employment status have changed since their cancer diagnosis.

DETAILED DESCRIPTION:
One in three breast cancer patients experiences treatment-related, cost-associated distress. This financial harm is termed "financial toxicity" (FT). FT is the strongest independent risk factor for diminished quality of life and patient-reported outcomes (PROs) among cancer patients. The present study will be the first prospective cohort study examining FT in breast cancer patients in Canada, or any other publicly-funded healthcare system.

The primary objective is to detect the prevalence and trajectory of FT using a validated instrument and its association with patient and treatment-related characteristics. The secondary objective is to assess the effects of financial toxicity on patient-reported quality of life, well-being, and satisfaction. The tertiary objective is to assess patients' baseline cost expectations for reconstructive surgery, actual out-of-pocket spending, private insurance or workplace benefits expenditure, and employment status, over the course of treatment.

Participants will be recruited at their consultation with the general surgeon, will consent to be observed for up to 1 year and be asked to complete a series of validated questionnaires, at baseline, 6 months, and 12 months.

The primary outcome is financial toxicity (FT), assessed using the COmprehensive Score for financial Toxicity (COST), a validated patient-reported outcome measure that uses a 12 item, five-point Likert scale type.

The secondary outcomes include (1) well-being and satisfaction, as measured by the BREAST-Q, (2) quality of life as measured by the 12-Item Short Form Health Survey (12-SF), (3) patient-level (age, co-morbidities, stage, socioeconomic status) and treatment-associated (complications, type of breast surgery, decision to have reconstruction, type of reconstruction), and (4) baseline cost expectations, out-of-pocket spending, private insurance or workplace benefits expenditure, and employment status, over the course of treatment.

Multivariate regression will be used to identify patient and treatment level factors associated with financial toxicity. First, the association between the COST scores and each survey question response, patient characteristic, and treatment factor will be determined. A stepwise linear regression will be completed with backward elimination to generate a list of co-variates based on their significance level. All variables in the final selected model has a significance level < 0.1. Other data will be characterized the study samples by presenting the means, standard deviations, and medians for continuous variables and frequencies for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Have an indication for surgical treatment of breast cancer
* 18 years of age or older
* Able to understand and communicate in English
* Have access to email and internet and are able to fill out an electronic survey

Exclusion Criteria:

- Patients will be excluded if they have recurrent or metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women undergoing surgery for breast cancer or risk reduction (e.g., BRCA) including both breast conservation or mastectomy, with or without reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Financial Toxicity (FT) | 12 months
  FT will be assessed using the COmprehensive Score for financial Toxicity (COST). The COST measure is an 11-item cancer-specific patient-reported outcome measure. Each item is scored on a 0 to 4-point Likert scale, where a lower total score represents greater financial distress.

SECONDARY OUTCOMES:
Financial Toxicity (FT) | Baseline, 6 months
  FT will be assessed using the COmprehensive Score for financial Toxicity (COST). The COST measure is an 11-item cancer-specific patient-reported outcome measure. Each item is scored on a 0 to 4-point Likert scale, where a lower total score represents greater financial distress.
Satisfaction with Breasts | Baseline, 6 months, 12 months
  This will be measured using the BREAST-Q questionnaire; Satisfaction with Breast Module. All questions are answered on Likert scales (scored 1-4). This module varies based on the type of breast surgery the patient underwent (mastectomy only, breast conserving surgery, or reconstruction). The answers of this section are totalled and compared to the equivalent Rasch transformed score. Zero represents the worst possible score and 100 represents the best.
Psychosocial Well-Being | Baseline, 6 months, 12 months
  This will be measured using the BREAST-Q questionnaire; Psychosocial Well-Being Module. All questions are answered on Likert scales (scored 1-5). The answers this section are totalled and compared to the equivalent Rasch transformed score. Zero represents the worst possible score and 100 represents the best.
Satisfaction with Surgeon | Baseline, 6 months, 12 months
  This will be measured using the BREAST-Q questionnaire; Satisfaction with Surgeon Module. All questions are answered on Likert scales (scored 0-4). The answers this section are totalled and compared to the equivalent Rasch transformed score. Zero represents the worst possible score and 100 represents the best.
Quality of Life (mental and physical health) | Baseline, 6 months, 12 months
  Quality of life, will be assessed using the 12-Item Short Form Health Survey (12-SF) that evaluates overall physical and mental health. The SF-12 is a general health patient-reported outcome measure that has 12 items, is reported 0 to 100 for two domains. Higher scores represent better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Coroneos, MD, MSc, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No